CLINICAL TRIAL: NCT04103853
Title: Safety, Tolerability, and Pharmacokinetics of Proxalutamide Therapy in Women With Metastatic Breast Cancer: an Open-label, Multi-center, Dose-escalating，Phase I/Ib Study.
Brief Title: Safety, Tolerability, and Pharmacokinetics of Proxalutamide Therapy in Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Sun Yat-sen University (Other); Ruijin Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Hebei Medical University Fourth Hospital (Other); Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT0918-CN-2001
Record Dates: First submitted 2019-09-20; First posted 2019-09-26 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Breast Cancer
Keywords: AR-positive metastatic breast cancer; Proxalutamide; metastatic breast cancer; GT0918
MeSH Terms: conditions — Breast Neoplasms | interventions — proxalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proxalutamide (Experimental): Stage one - Dose climbing:
  Each dose cohort will assess toxicity within the 35 days following the first dose of GT0918.
  Stage two- the expansion cohort :
  30 patients will be enrolled to the 200mg cohort . 15 patients will be enrolled to the 300mg cohort.
  Interventions: Drug: Proxalutamide

INTERVENTIONS:
Drug: Proxalutamide — Stage1:Dose esclation. Stage2:the expansion cohort where one or no DLT takes place in planned study cohort.

SUMMARY:
This study is a multi-center, open-label, dose-esclation I/Ib clinical study to explore safety, efficacy an pharmacokinetics of proxalutamide in patients with metastatic breast cancer.

This study includes two stages, stage I: single- and multiple-dose tolerance and pharmacokinetic study; stage 2: preliminary efficacy and safety study.

DETAILED DESCRIPTION:
This study is a multi-center, open-label, dose-esclation study.

Subjects will be enrolled to the 100mg, 200mg, 300mg, 400mg and 500mg group in turn. Unless DLT was found, the dose esclation will continue. 28 days of DLT observation period is needed after 7-day single dose administration, until disease progression, intolerable toxicities (AEs), or withdrawn consent.

After the completion of stage 1, 2 doses for the stage 2 will be determined. In stage 2, patients with AR-positive metastatic breast cancer will be selected to explore the efficacy and safety of proxalutamide, and biomarkers will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years female;
2. Stage 1:Histology or cytology confirmed metastatic breast cancer, first-line chemotherapy or targeted therapy failure or intolerance

   Stage 2: Histological or cytological confirmed metastatic breast cancer patients who failed or intolerant to anti-tumor therapy; have a positive AR test result;
3. At least one measurable lesion based on RECIST version 1.1 ;
4. ECOG performance status: 0-1;
5. Have a predicted life expectancy of greater than 3 months;
6. The functions of the important organs are confirmed with the following requirement:

   * Hemoglobin (HGB) ≥ 90 g/L(no blood transfusion within 14 days );
   * Absolute neutrophil count (ANC) ≥ 1.5×10^9/L；
   * Platelets (PLT) ≥ 100×10^9/L(If the coagulation function is normal,Platelets (PLT) ≥ 75×10^9/L )；
   * Total bilirubin (TBIL) ≤ 1.5× Upper limit of normal value (ULN) -Aspartate aminotransferase (AST), alkaline phosphatase (ALP), and alanine -
   * Aminotransferase (ALT) ≤2.5× ULN
7. Understand and voluntarily sign the informed consent form；
8. Subject is willing and able to comply with all protocol required visits and assessments；

Exclusion Criteria:

1. Pregnant, lactating women, or those who have fertility and are reluctant to take effective contraceptive measures;
2. Prior chemotherapy, radiation, targeted therapy ,androgen receptor inhibitors therapy (abiraterone,enzalutamide,etc )，other endocrine therapy ，and has acceptted traditional chinese herbal medicine treatment less than 4 weeks prior to the start of study medication.
3. Has severe cardiovascular disease
4. The toxicity of the previous treatment plan has not been restored before enrollment, and there is still non-hematologic toxicity of grade 1 or above (except for hair loss)
5. Known gastrointestinal disease or condition that affects the absorption of GT0918;
6. Known or suspected brain metastases, including the central nervous system and spinal cord compression or meningeal metastasis;
7. History of severe central nervous system diseases (including patients with epilepsy);
8. Known hypersensitivity to proxalutmide or its excipients.
9. Participated in clinical trials of other drugs or medical devices within one month prior to screening, or plan to participate in any other clinical trials during the study period;
10. Subjects with any other serious disease considered by the investigator not in the condition to enter into the trial;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicity(DLT) | 35 days
  Each dose cohort will initially include 3 evaluable patients for assessment of toxicity within the 35 days following the first dose of GT0918.
maximum tolerated dose (MTD) | 35 days
  100 mg, 200 mg, 300 mg, 400 mg or 500 mg of GT0918
Disease Control Rate(DCR) | 16 weeks
  Preliminary evaluation of the DCR of GT0918 tablets in AR positive metastatic breast cancer patients, and determination of the recommended dose of proclamine in clinical trials.

SECONDARY OUTCOMES:
maximum concentration (Cmax) | 35 days
  Pharmacokinetics
time that maximum concentration is observed (tmax) | 35 days
  Pharmacokinetics
area under the concentration time-curve from time zero to infinity (AUC0∞) | 35 days
  Pharmacokinetics
terminal elimination half life (t½) | 35 days
  Pharmacokinetics
drug clearance (CL) | 35 days
  Pharmacokinetics
apparent volume of distribution (Vd) | 35 days
  Pharmacokinetics
Number of participants with treatment-related adverse events as assessed by CTCAE V4.03 | 16 weeks
  200 mg, 300 mg of GT0918

CONTACTS AND LOCATIONS:
Overall Officials: Ke Chen, Study Director — Suzhou Kintor Pharmaceuticals,inc
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun-Yat-sen University Cancer center, Guangzhou, Fujian
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang H, Ouyang Q, Yin Y, Tong Z, Shen K, Yuan Z, Geng C, Liu Y, Song G, Ran R, Li W, Qu Q, Wang M, Meng L, Tong Y, Li H. Proxalutamide in patients with AR-positive metastatic breast cancer: Results from an open-label multicentre phase Ib study and biomarker analysis. Eur J Cancer. 2022 Nov;176:1-12. doi: 10.1016/j.ejca.2022.08.025. Epub 2022 Sep 28. PMID 36182805
- [Derived] Li H, Song G, Zhou Q, Ran R, Jiang H, Zhang R, Liu Y, Zhang J, Meng L, Ma L, Sun Y, Wang M, Zhou Q, Yan H, Zhou Q, Dong X, Tong Y. Activity of preclinical and phase I clinical trial of a novel androgen receptor antagonist GT0918 in metastatic breast cancer. Breast Cancer Res Treat. 2021 Oct;189(3):725-736. doi: 10.1007/s10549-021-06345-x. Epub 2021 Aug 14. PMID 34392453